CLINICAL TRIAL: NCT04328051
Title: Influence of the Implant-prosthetic Connection in the Marginal Bone Loss and Bacterial Leakage. A Randomized Controlled Trial
Brief Title: Influence of the Implant-prosthetic Connection in the Marginal Bone Loss and Bacterial Leakage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Octavi Camps-Font, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBarcelonaOralSurgery2
Record Dates: First submitted 2018-06-21; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Dental Implant; Bone Loss; Bacterial Infections
Keywords: Dental Implant; Internal Connection; External Connection; Conical Connection; Marginal Bone Loss; Implant Prosthetic Connection; Bacterial Leakage
MeSH Terms: conditions — Bone Diseases, Metabolic; Bacterial Infections | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Active comparator: Ocean E.C.®, Avinent Implant System S.L., Santpedor, Spain. Active comparator: Ocean I.C.®, Avinent Implant System S.L., Santpedor, Spain. Active comparator: Ocean C.C.®, Avinent Implant System S.L., Santpedor, Spain.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will not know the type of connection of his or her implant until the study has finished. Outcome Assessor will be blinded. In the radiographic evaluation the implant-abutment connection will be hidden to assess the marginal bone loss.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ocean E.C.®, Avinent Implant System S.L. (Active Comparator): Dental implant with geometry adapted to the biologic architecture of the bone, with platform switching with a positive angle and machined surface with micro-threads in the cervical region. Asymmetric and progressive threads in its body with a double thread pitch. Point-ratio geometry on its apical region, Biomimetic Advanced Surface and external hexagon connection.
  Interventions: Other: Dental Implant Placement
- Ocean I.C.®, Avinent Implant System S.L. (Active Comparator): Dental implant with geometry adapted to the biologic architecture of the bone, with platform switching with a positive angle and machined surface with micro-threads in the cervical region. Asymmetric and progressive threads in its body with a double thread pitch. Point-ratio geometry on its apical region, Biomimetic Advanced Surface and internal hexagon connection.
  Interventions: Other: Dental Implant Placement
- Ocean C.C.®, Avinent Implant System S.L. (Active Comparator): Dental implant with geometry adapted to the biologic architecture of the bone, with platform switching with a positive angle and machined surface with micro-threads in the cervical region. Asymmetric and progressive threads in its body with a double thread pitch. Point-ratio geometry on its apical region, Biomimetic Advanced Surface and conical connection.
  Interventions: Other: Dental Implant Placement

INTERVENTIONS:
Other: Dental Implant Placement — Antibiotic prophylaxis will be done. After rinsing with 0.12 % chlorhexidine, patients will receive local anaesthesia. A crestal incision will be done and a mucoperiostic flap will be raised. As the commercial specifies, progressive diameter drills will be used under constant sterile saline irrigation to prepare the implant site. Once finished the drilling sequence, one investigator will open the opaque envelope to know which type of implant, depending on the connection, has to be placed by the surgeon. Dental implant will be placed crestally and depending if it has primary stability or not, it will be leaded submerged or non-submerged. The flap will be repositioned and sutured without tension with 4/0 polyamide. Postoperative instructions and medication will be prescribed and explained.
  Other Names: Surgery

SUMMARY:
This study consists in a double-blinded randomized controlled trial which objective is to assess the effect of the implant-abutment connection type -external hexagon, internal hexagon and conical connection- in the periimplant marginal bone loss in vertical side and the bacterial leakage 12 months after prosthesis placement.

DETAILED DESCRIPTION:
Location: This study is going to take place in the Dentistry Hospital of the University of Barcelona (Campus of Bellvitge).

Study subjects: The sample (105 patients) consists of patients with single tooth edentulous spaces or posterior maxillary and/or mandible edentulous spaces in need of dental implants with screw-retained single fixed crowns. All of them are being properly informed about the study according to the Comité Ético (CEIC) del Hospital Odontològic Universitat de Barcelona guidelines, and informed consent must be signed prior to the interventions.

Material: Registration papers for the study, dental implants, surgery material, prosthetic components, Florida Probe Software®, Periapical x-rays, computer, Software Stata 14 and Software ImageJ®.

Determinations: Clinical, radiographic and microbiologic measures since implant placement, prosthesis placement and 3, 6, 9 and 12 months after it.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who accept signing voluntarily the informed consent before doing any action related to the study.
* ≥18-years-old patients.
* Edentulous single spaces or edentulous posterior maxilla or mandible (from the first premolar to the second molar) with screw-retained single fixed crowns.
* Single implants successfully osseointegrated placed at least 16 weeks post-extraction.
* O'Leary plaque index and or bleeding on probing ≤25%.
* Dental implants with screwed-retained prosthesis.

Exclusion Criteria:

* Systemic diseases that can interfere dental implant placement.
* Any contraindication for surgery procedures.
* Heavy smokers (> 20cig/day).
* Background of drug abuse or other factors such as psychiatric diseases that, in opinion of the examiner, could interfere with the ability of the patient to cooperate and compliment with the study.
* Patients who have had participated with another clinical trial the last 30 days.
* Pregnant women or in lactation.
* Patients with bad oral hygiene or not motivated.
* Probing pockets depths with bleeding of ≥4 mm on a tooth adjacent to the edentulous space.
* Guided bone regeneration required in the same time of the implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-06-13 (Estimated); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
Change in Vertical Marginal Bone Loss (VMBL) | Since implant placement (Timing 0) through study completion (Timing 5), an average of 1 year.
  Distance in millimetres between the implant platform and the point of the intra-bone defect that is more apical.

SECONDARY OUTCOMES:
Vertical Marginal Bone Loss Tax | 12 months after prosthesis placement.
  Vertical bone loss in millimetres per implant and unit of time.
Early implant failure | Since implant placement (Timing 0) through prosthesis placement (Timing 1).
  Implant with mobility or failure of the osseointegration process before the prosthesis placement.
Late implant failure | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Implant with mobility or failure of the osseointegration process after the prosthesis placement.
Probing pocket depth | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Distance in millimetres from the gingival margin to the bottom of the periodontal pocket measured with the periodontal probe. Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal).
Mucosal recession | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Distance in millimetres from the cemento-enamel junction of the tooth or from the implant platform to the gingival margin when it is located apically. Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal).
Mucosal hyperplasia | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Distance in millimetres from the gingival margin to the cemento-enamel junction of the tooth or to the implant platform when the gingiva is located more coronal than them. Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal).
Clinical attachment level | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Probing pocket depth (mm) plus the recession (mm) or probing pocket depth minus the hyperplasia (mm). Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal).
O'Leary plaque index | First visit
  Plaque presence in the dentogingival or implantogingival union. Determined in four points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual). Expressed as the percentage (%) of tooth or implant surfaces with plaque presence divided with the total of tooth or implant surfaces in mouth and multiplied per 100.
Bleeding on probing | Since first visit through study completion (Timing 5), an average of 1 year.
  Presence of blood in the gingival margin after determining the probing pocket depth. Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal). Expressed as the percentage (%) of tooth or implant surfaces with blood divided with the total of tooth or implant surfaces in mouth and multiplied per 100.
Suppuration on probing | Since first visit through study completion (Timing 5), an average of 1 year.
  Presence of purulent material in the gingival margin after determining the probing pocket depth. Determined in six points per tooth or implant (Buccal: mesial, medial and distal. Palatal or lingual: mesial, medial and distal). Expressed as the percentage (%) of tooth or implant surfaces with pus divided with the total of tooth or implant surfaces in mouth and multiplied per 100.
Prosthetic complications | Since prosthesis placement (Timing 1) through study completion (Timing 5), an average of 1 year.
  Screw (which connects the crown with the implant) fracture or prosthesis fracture, chipping of the ceramic prosthesis, loosening of the screw (which connects the crown with the implant) or any other prosthetic components.
Bacterial leakage | 12 months after prosthesis placement.
  Quantitative PCR in real time to determine the total amount of bacteria and in particular, of 10 pathogenic species: Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythensis, Treponema denticola, Prevotella intermedia, Peptostreptococcus micros, Fusobacterium nucleatum, Campylobacter rectus, Eikenella corrodens and Candida albicans.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Figueiredo, DDS, MS, PhD, Study Director — University of Barcelona; Eduard Valmaseda-Castellón, DDS, MS, PhD, Study Chair — University of Barcelona; Octavi Camps-Font, DDS, MS, Principal Investigator — University of Barcelona; Roxana Ghiorghiu, DDS, MS, Principal Investigator — University of Barcelona; Laura Rubianes-Porta, DDS, MS, Principal Investigator — University of Barcelona; Anna Piñol-Olea, DDS, MS, Principal Investigator — University of Barcelona
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Under request

REFERENCES:
- [Background] Branemark PI, Adell R, Breine U, Hansson BO, Lindstrom J, Ohlsson A. Intra-osseous anchorage of dental prostheses. I. Experimental studies. Scand J Plast Reconstr Surg. 1969;3(2):81-100. doi: 10.3109/02844316909036699. No abstract available. PMID 4924041
- [Background] Albrektsson T, Donos N; Working Group 1. Implant survival and complications. The Third EAO consensus conference 2012. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:63-5. doi: 10.1111/j.1600-0501.2012.02557.x. PMID 23062128
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Buser D, Ingimarsson S, Dula K, Lussi A, Hirt HP, Belser UC. Long-term stability of osseointegrated implants in augmented bone: a 5-year prospective study in partially edentulous patients. Int J Periodontics Restorative Dent. 2002 Apr;22(2):109-17. PMID 12019706
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Oh TJ, Yoon J, Misch CE, Wang HL. The causes of early implant bone loss: myth or science? J Periodontol. 2002 Mar;73(3):322-33. doi: 10.1902/jop.2002.73.3.322. PMID 11922263
- [Background] Quirynen M, Naert I, van Steenberghe D. Fixture design and overload influence marginal bone loss and fixture success in the Branemark system. Clin Oral Implants Res. 1992 Sep;3(3):104-11. doi: 10.1034/j.1600-0501.1992.030302.x. PMID 1290790
- [Background] Malevez C, Hermans M, Daelemans P. Marginal bone levels at Branemark system implants used for single tooth restoration. The influence of implant design and anatomical region. Clin Oral Implants Res. 1996 Jun;7(2):162-9. doi: 10.1034/j.1600-0501.1996.070210.x. PMID 9002835
- [Background] Vidyasagar L, Apse P. Dental implant design and biological effects on bone implant interface. Baltic Dent Maxillofac J. 2004;6:51-4.
- [Background] Isidor F. Influence of forces on peri-implant bone. Clin Oral Implants Res. 2006 Oct;17 Suppl 2:8-18. doi: 10.1111/j.1600-0501.2006.01360.x. PMID 16968378
- [Background] Abrahamsson I, Berglundh T. Effects of different implant surfaces and designs on marginal bone-level alterations: a review. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:207-15. doi: 10.1111/j.1600-0501.2009.01783.x. PMID 19663966
- [Background] Koo KT, Lee EJ, Kim JY, Seol YJ, Han JS, Kim TI, Lee YM, Ku Y, Wikesjo UM, Rhyu IC. The effect of internal versus external abutment connection modes on crestal bone changes around dental implants: a radiographic analysis. J Periodontol. 2012 Sep;83(9):1104-9. doi: 10.1902/jop.2011.110456. Epub 2011 Dec 6. PMID 22145806
- [Background] Nishioka RS, de Vasconcellos LG, de Melo Nishioka GN. Comparative strain gauge analysis of external and internal hexagon, Morse taper, and influence of straight and offset implant configuration. Implant Dent. 2011 Apr;20(2):e24-32. doi: 10.1097/ID.0b013e318211fce8. PMID 21448016
- [Background] Lin MI, Shen YW, Huang HL, Hsu JT, Fuh LJ. A retrospective study of implant-abutment connections on crestal bone level. J Dent Res. 2013 Dec;92(12 Suppl):202S-7S. doi: 10.1177/0022034513510322. Epub 2013 Oct 24. PMID 24158343
- [Background] Astrand P, Engquist B, Dahlgren S, Grondahl K, Engquist E, Feldmann H. Astra Tech and Branemark system implants: a 5-year prospective study of marginal bone reactions. Clin Oral Implants Res. 2004 Aug;15(4):413-20. doi: 10.1111/j.1600-0501.2004.01028.x. PMID 15248875